CLINICAL TRIAL: NCT05841329
Title: Efficacy of tDCS to Enhance Virtual Reality Exposure Therapy Response in Acrophobia: A Randomized Controlled Trial
Brief Title: Efficacy of tDCS to Enhance Virtual Reality Exposure Therapy Response in Acrophobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMHC-VR-001
Record Dates: First submitted 2023-03-11; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-03

CONDITIONS: Acrophobia; Transcranial Direct Current Stimulation
Keywords: virtual reality exposure therapy; acrophobia; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Acrophobia | interventions — Transcranial Direct Current Stimulation; Virtual Reality Exposure Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active group (Active Comparator): receive active tDCS before VRET
  Interventions: Device: tDCS; Behavioral: virtual reality exposure therapy
- sham group (Sham Comparator): receive sham tDCS before VRET
  Interventions: Behavioral: virtual reality exposure therapy

INTERVENTIONS:
Device: tDCS — High-definition tDCS (HD-tDCS, 4×1 montage, with 1 anode and 4 cathodes, (Soterix Medical, New York, NY, USA) was applied with battery-driven electrical stimulator (2001&4×1-C3A). The center electrode was anode and placed over FPz (according to the EEG 10-20 system in order to target the medial prefrontal cortex). The reference electrodes were cathodes and placed over AF7, AF8, F3, F4(see fig. 3). Participants were randomized to receive 20 minutes of active(1.5mA) or sham (0 mA) tDCS in a single-blind design. In order to ensure that participants can gradually adapted to the current change, there was a 15-second current rising process before the stimulation and, a 15-second current falling process after the stimulation. For sham tDCS, the device was automatically turned off after current reached 1.5 mA, thus providing 30s of ramping current stimulation, which made it difficult for participants to distinguish which kinds of stimulation they received.
  Arms: active group
Behavioral: virtual reality exposure therapy — The VRET was adapted on the basis of Öst's single exposure treatment paradigm and conducted by experienced psychotherapists following a standard exposure treatment manual.. An exposure therapy was divided into three parts: psychological education, exposure intervention and summary. Each scene started with a 10-min psychological education followed up with the tDCS stimulation. In exposure trail, participants ought to take an elevator to 100th, observe the environment and look down on the platform. The psychotherapist guided participants to be exposed to the VR environment and helped them experience the process of anxiety decline in the exposure trail.

SUMMARY:
The goal of this clinical trial is to examine whether transcranial direct current stimulation(tDCS) can enhance the effect of virtual reality exposure therapy(VRET) in acrophobia in college students with significant fear of heights. The main question it aims to answer are:

• the enhancement of tDCS on the effect of VRET Participants will randomly allocated to tDCS active stimulated group and sham stimulated group and receive VRET.

ELIGIBILITY:
Inclusion Criteria:

* the score of the AQ-Anxiety had to be at least 45.45(1SD below the mean of a previous acrophobia sample(Cohen, 1977));
* the participants had the avoidance behaviors in daily life and recognized the fear of height was excessive and unnecessary (the severity of fear of heights not less than 5 points at a scale from 0 to 10).

Exclusion Criteria:

* previous treatment for acrophobia, history or family history of any mental disorder (except for acrophobia), metal parts in the head, medical implants, increased intracranial pressure, pregnancy, current involvement in psycho- or pharmacotherapy, and cardiovascular or neurological diseases.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Acrophobia Questionnaire(AQ) | one day(baseline, after invervention)
  It consists of two scales that assess fear (Anxiety, ranging from 0 to 120, involving 20 height situations scored on a seven-point Likert scale; Cronbach' α = 0.80) and avoidance behaviors (Avoidance, ranging from 0 to 40, involving 20 height situations scored on a three-point Likert scale; Cronbach' α = 0.70) of height. Each scale contains 20 scenarios about height situation, such as "Standing next to an open window on the third floor". AQ is widely used to measure fear of heights and has good reliability.
  Change from Baseline AQ at post-intervention was assessed in the study.

SECONDARY OUTCOMES:
Heights Interpretation Questionnaire(HIQ) | one day(baseline, after invervention)
  This scale is a 16-item self-report questionnaire that are rated on a 5-point Likert scale(1 to 5). It was designed to measure height-relevant interpretations. Total scores range from 16 to 80, with higher scores indicating more height-relevant interpretations.
  Change from Baseline HIQ at post-intervention was assessed in the study.
State-Trait Anxiety Inventory Form Y, (STAI-Y) | one day(baseline, after invervention)
  This scale is a 40-item self-report questionnaire that are rated on a 4-point Likert scale(1 to 4). Higher scores indicate more state and trait anxiety.
  Change from Baseline STAI-Y at post-intervention was assessed in the study.
the Beck Anxiety Inventory(BAI) | one day(baseline, after invervention)
  It is an inventory of anxiety symptoms with 18 items that are rated on a 5-point Likert scale(0 to 4). Total scores range from 0 to 72, with higher scores indicating more severe anxiety symptoms.
  Change from Baseline BAI at post-intervention was assessed in the study.
Subjective Units of Distress Scale(SUDS) | assessed every five minutes during intervention
  This scale is used to assess the level of anxiety with 10 items that are rated from 0-10 point. The higher score indicates more severe current anxiety or distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No